CLINICAL TRIAL: NCT04750512
Title: Comparing Erector Spinae Plane (ESP) and Transversus Abdominis Plane (TAP) Block Analgesic Effect After Robotic TAPP Abdominal Hernia Repair: a Single Center, Randomized, Triple-blind, Controlled Trial
Brief Title: Comparing Erector Spinae Plane (ESP) and Transversus Abdominis Plane (TAP) Block in Inguinal Hernia
Acronym: TAPESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ghielmini Enea (Other)
Responsible Party: Sponsor-Investigator, Ghielmini Enea, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORBV - CHIR - TAPESP
Record Dates: First submitted 2021-02-09; First posted 2021-02-11 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Inguinal Hernia; Postoperative Pain; Anesthesia, Local; Anesthesia Complication
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is a single center, prospective, randomized, "double-dummy" placebo-blinded, controlled superiority trial in 2 parallel arms comparing the efficacy and safety of the ESP Block and the TAP block on patients undergoing elective robot-assisted inguinal hernia repair.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: According to the randomization arm patients will receive:
  * sham US-guided ESP block + US-guided TAP block before laparoscopic hernia repair
  * US-guided ESP block + sham US-guided TAP block before laparoscopic hernia repair Allocation will take place immediately before the intervention by the means of access to centralized, real-time allocation through a computer program.
  Personnel not directly involved with patient care will prepare a saline solution and a ropivacaine solution which will be allocated respectively to ESP or TAP block according to randomization.
  This will allow blinding of patients, care providers and data collectors. Analysis will be done on allocation-concealed data, permitting blinded analysis.
  Unbliding will be permitted if by doing so harm to one or more patients can be avoided or treated. After information of one of the principal investigators, specific patient allocation will be retrieved from the randomization program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real ESP, placebo TAP (Experimental): US-guided ESP block + sham US-guided TAP block
  Interventions: Procedure: ESP block
- real TAP, placebo ESP (Active Comparator): sham US-guided ESP block + US-guided TAP block before laparoscopic hernia repair
  Interventions: Procedure: TAP block

INTERVENTIONS:
Procedure: ESP block — US guided ESP infiltration (saline solution vs Ropivacaine 0.2% according to randomization): bilateral injection of 30ml (60ml total) under US guidance between the deep fascia of erector spinae muscle and the the two transverse process at the level of the 10th thoracic vertebrae
  Arms: real ESP, placebo TAP
Procedure: TAP block — US guided TAP block (saline solution vs Ropivacaine 0.2% according to randomization):
  bilateral injection of 30ml (total 60ml) under US guidance in the plane between the internal oblique and transversus abdominis muscles at the level of the midaxillary line in the Petit triangle.
  Arms: real TAP, placebo ESP

SUMMARY:
The Erectore Spinae Plane Block (ESP Block) is a recently described technique for regional anesthesia that has shown promising results in the treatment of pain after thoracic surgery. It involves the injection of local anesthetic behind the musculature of the back.

The investigators intend to compare this technique with a more standardized one, the TAP Block, which involves injection of anesthetic behind the musculature of the abdomen.

50 patients undergoing robotic inguinal hernia repair under general anesthesia will be randomly selected to receive, in addition to general anesthesia, either the ESP block or the TAP block. Patients receiving an ESP Block will also receive an injection of saline solution in the TAP injection site, and the other way around. This will prevent preconceived ideas on either technique to influence the evaluationso of the effect.

Pain scores and consumption of pain medication will be recorded during the 24 hours following the operation to compare the effect of the two techniques.

DETAILED DESCRIPTION:
In the recent era of increased awareness towards the risks and complications of opioid treatment, pain management after common surgical interventions by the means of regional anesthesia is of renewed interest for both clinical and logistic reasons, as it is known that good pain management reduces complications and cost associated to surgery.

Regional and local anesthetic techniques after inguinal hernia surgery have been the topic of multiple studies, comparing various infiltrative methods, including wound infiltration, port site infiltration, iliohypogastric and ilioinguinal nerve block, paravertebral and transversus abdominis plane (TAP) block and epidural analgesia. Most methods investigate pain treatment in the setting of open surgery. The progressive evolution towards laparoscopic and robot-assisted methods changes the mechanisms of surgical pain and, with it, the rational for the choice of the analgesic technique adopted. The transversus abdominis plane (TAP) has become a widely used technique and has been demonstrated to be associated to a mild opioid sparing effect, but with inconsistent results.

The erector spinae plane block is a promising technique, recently described and used especially in thoracic surgery. Multiple case reports and studies in pediatrics report it to be a safe and effective method for abdominal surgery as well, but no prospective randomized trials were published to date in the adult population, particularly with regard to laparoscopic or robotic hernia repair. A prospective comparison between the two techniques is therefore needed in this specific context.

Hypothesis and primary objective:

The investigators hypothesize the superiority of the ESP-block to the TAP-block with respect to post-operative pain control after abdominal surgery, leading to a reduction in reserve analgesic consumption.

Our objective is to compare the clinical outcomes and safety of ESP block versus TAP block in patients undergoing robot-assisted TAPP inguinal hernia repair.

Primary and secondary endpoints:

Primary Endpoint:

* The highest VAS score reported between end of sedation and 6 hours after surgery or discharge of the patient, whichever comes first Secondary Endpoints
* Time to first rescue analgesic
* Total dose of rescue opioids (morphine equiavalents) in the first 24 hours after surgery
* Time of first walk after surgery
* Need for anti-nausea medication (dosage, doses and time points)
* Episodes of vomiting
* Episodes of urinary retention
* Patient's satisfaction (measured on the validated LPPS questionnaire for the perioperative patients' satisfaction )
* Length of hospital stay

Study design This is a single center, prospective, randomized, placebo-blinded, controlled superiority trial in 2 parallel arms comparing the efficacy and safety of the ESP Block and the TAP block on patients undergoing elective robot-assisted inguinal hernia repair.

Follow up will consist in the hospitalization period plus one telephone consultation at 24 hours after hospitalization.

Methods of minimizing bias:

Randomisation - Patients will be randomized in a 1:1 ratio by a computer generated random number sequence through the RedCap software system.

Blinding procedures

According to the randomization arm patients will receive:

* sham US-guided ESP block + US-guided TAP block before laparoscopic hernia repair
* US-guided ESP block + sham US-guided TAP block before laparoscopic hernia repair Allocation will take place immediately before the intervention by the means of access to centralized, real-time allocation through a computer program.

Personnel not directly involved with patient care will prepare a saline solution and a ropivacaine solution which will be allocated respectively to ESP or TAP block according to randomization.

This will allow blinding of patients, care providers and data collectors. Analysis will be done on allocation-concealed data, permitting blinded analysis.

Unbliding will be permitted if by doing so harm to one or more patients can be avoided or treated. After information of one of the principal investigators, specific patient allocation will be retrieved from the randomization program.

Other methods of minimising bias

Pain scores will be measured at 1, 3, 6, 12 and 24 hours after extubation and at the time of administration of reserve analgesics.

The administration of reserve analgesics will follow a standardized internal protocol.

Questionnaires validated to assess functional results after hernia surgery will be used for this study:

* pain: Visual Analogue Scale (VAS)
* surgical complications classification: Clavien Dindo's classification
* comorbidities : American Society of Anesthesiology (ASA) score
* validated LPPS questionnaire for the perioperative patients' satisfaction [21]
* EHS inguinal hernia classification

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Patients over 18 years of age
* Planned elective unilateral or bilateral robot-assisted TAPP hernia repair, with mesh placement

Exclusion Criteria:

* Contraindications to ropivacaine or opioids, e.g. known hypersensitivity or allergy
* Infections at the injection site
* Coagulopathies or ongoing anticoagulant therapy
* Concomitant surgery other than inguinal or umbilical hernia repair
* Pre-operative chronic narcotic usage
* Known chronic pain syndrome
* Prior complex abdominal wall reconstruction
* Frail patients for whom a prolonged sedation can be detrimental
* Women who are pregnant
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to consent or follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Highest Visual Analogue Scale | Between end of sedation and 6 hours after surgery
  0 to 100mm, highest equals to more pain

SECONDARY OUTCOMES:
Visual Analogue Scale score at rest and at movement | 1, 3, 6, 12 and 24 hours after surgery
  0 to 100mm, highest equals to more pain
Total dose of rescue opioids | in the first 24 hours after surgery
  (morphine equiavalents)
Time of first walk after surgery | 24 hours
Episodes of urinary retention | 24 hours
Need for anti-nausea medication (dosage, doses and time points) | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- ORBV, Bellinzona, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ghielmini EM, Greco L, Spampatti S, Kubli R, Saporito A, La Regina D. Erector Spinae Plane Block versus Transversus Abdominis Plane Block for Robotic Inguinal Hernia Repair: A Blinded, Active-Controlled, Randomized Trial. Pain Physician. 2024 Jan;27(1):27-34. PMID 38285028